CLINICAL TRIAL: NCT06557473
Title: Hemodynamic Stability of Fentanyl Based Versus Lidocaine Based Induction of Anesthesia in Hypertensive Adults
Brief Title: Lidocaine Versus Fentanyl for Hemodynamic Stability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Moshira sayed mohamed, lecturer, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT (812)
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Hypertension; Fentanyl; Lidocaine
Keywords: Hypertension; Postinduction hypotension; Lidocaine; Fentanyl
MeSH Terms: conditions — Hypertension | interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: comparison of lidocaine and fentanyl in hemodynamic stability after induction of general anesthesia in hypertensive patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An investigator not participating in the study was responsible for drug preparation and allocation according the computer generated random numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The lidocaine group (Active Comparator): Anesthesia will be induced using 1.5 mg/kg lidocaine in the lidocaine group (L), 2mg/kg propofol, and 0.5 mg atracurium.
  Interventions: Drug: Lidocaine IV
- The fentanyl group (Placebo Comparator): Anesthesia will be induced using 2 µg/kg fentanyl in the fentanyl group (F), 2mg/kg propofol, and 0.5 mg atracurium.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Lidocaine IV — 1.5mg/kg IV for induction of GA
  Arms: The lidocaine group
Drug: Fentanyl — Fentanyl IV 2 µg/kg for GA induction
  Arms: The fentanyl group

SUMMARY:
Hypertension is an important health challenge that affects millions of people across the world today and is a major risk factor for multiple system comorbidities. Intraoperative hypotension may lead to negative outcomes. 'Post-induction hypotension' (PIH; i.e. arterial hypotension defined as hypotension during the first 20 min after anesthesia induction, or from anesthesia induction until the beginning of surgery) and 'early intraoperative hypotension' (eIOH; i.e. arterial hypotension occurring during the first 30 min of surgery). Lidocaine is a local anesthetic drug with multiple systemic uses. Systemic lidocaine used as at the perioperative period has analgesic, and anti-inflammatory properties which make it capable of reducing intra- and postoperative drug consumptions and patients' hospital stay. Therefore, we hypothesize that the use of lidocaine as an adjuvant to propofol might reduce the risk of post induction hypotension and hence having more stable hemodynamic profile during induction of anesthesia.

DETAILED DESCRIPTION:
Since post induction hypotension is mainly caused by anesthetic drugs, developing a technique for the induction of anesthesia that provides adequate hypnosis with stable hemodynamics during surgery is critical, especially for hypertensive patients. (4) Propofol is the most commonly used drug for anesthesia induction; however, its use is usually associated with hypotension through vasodilation and direct myocardial depression. (5) Opioid drugs are usually added to propofol to potentiate its hypnotic effect; however, they also potentiate propofol's negative hemodynamic effect at the same degree, even with low doses of propofol (5).

Lidocaine is a local anesthetic drug with multiple systemic uses. Systemic lidocaine used as at the perioperative period has analgesic, and anti-inflammatory properties which make it capable of reducing intra- and postoperative drug consumptions and patients' hospital stay. (6) Lidocaine/ketamine combination showed a favorable hemodynamic profile following rapid-sequence induction of anesthesia in septic shock patients [14]. Therefore, we hypothesize that the use of lidocaine as an adjuvant to propofol might reduce the risk of post induction hypotension and hence having more stable hemodynamic profile during induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. ASA II, Hypertensive patients with the following criteria:

   * Diagnosed with hypertension more than 5 years and on continuous medications.
   * Controlled hypertension (systolic pressure < 140 mm Hg and the diastolic < 90 mm Hg).
2. Age: 18-60 years of both sexes.
3. Elective non cardiac surgery requiring general anesthesia.

Exclusion Criteria:

1. Uncontrolled hypertension (SPB > 140 mm Hg) OR (DBP < 90 mm HG).
2. SVV (stroke volume variability) ≥ 13.
3. Patients with suspected difficult intubation as judged by the attending anesthetist during the preoperative assessment and patients for whom an alternative device other than an endotracheal tube will be considered.
4. Pregnancy.
5. History of drug abuse.
6. Obese patients (BMI ≥ 35kg/m2).
7. Allergy to any of the used medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
MAP | 1 minute after GA induction
  Mean Arterial blood pressure 1 minute after induction of anesthesia.

SECONDARY OUTCOMES:
Number of hypotensive episodes | 20 minutes
  MAP less than 65 mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be available upon request from the principal investigator

REFERENCES:
- [Background] Yancey R. Anesthetic Management of the Hypertensive Patient: Part II. Anesth Prog. 2018 Fall;65(3):206-213. doi: 10.2344/anpr-65-03-17. PMID 30235430
- [Background] Aissaoui Y, Jozwiak M, Bahi M, Belhadj A, Alaoui H, Qamous Y, Serghini I, Seddiki R. Prediction of post-induction hypotension by point-of-care echocardiography: A prospective observational study. Anaesth Crit Care Pain Med. 2022 Aug;41(4):101090. doi: 10.1016/j.accpm.2022.101090. Epub 2022 May 1. PMID 35508291
- [Background] Hu AM, Qiu Y, Zhang P, Zhao R, Li ST, Zhang YX, Zheng ZH, Hu BL, Yang YL, Zhang ZJ. Higher versus lower mean arterial pressure target management in older patients having non-cardiothoracic surgery: A prospective randomized controlled trial. J Clin Anesth. 2021 May;69:110150. doi: 10.1016/j.jclinane.2020.110150. Epub 2021 Jan 6. PMID 33418429